CLINICAL TRIAL: NCT06355349
Title: A Randomized, Open-label, Single Dose, 2x4 Crossover Study to Evaluate the Safety and Pharmacokinetic Characteristics After Co-administration of JW0101 and C2101 and Administration of JW0102 in Healthy Volunteers Under Fasting Conditions
Brief Title: To Evaluate the Safety and PK Characteristics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: JW22101
Record Dates: First submitted 2024-03-29; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Other): Treatment A: Co-administration of 1 tablet of JW0101 and 1 tablet of C2101 Treatment B: Administration alone of 1 tablet of JW0102
  Tablet, Oral, QD for 1 Day, Washout period is more than 21 days after administration
  Interventions: Drug: Reference Drug or Test Drug
- Sequence B (Other): Treatment A: Co-administration of 1 tablet of JW0101 and 1 tablet of C2101 Treatment B: Administration alone of 1 tablet of JW0102
  Tablet, Oral, QD for 1 Day, Washout period is more than 21 days after administration
  Interventions: Drug: Reference Drug or Test Drug

INTERVENTIONS:
Drug: Reference Drug or Test Drug — Tablet, Oral, QD for 1 Day, Washout period is more than 21 days after administration
  Other Names: Reference Drug(JW0101 and C2101) or Test Drug(JW0102)

SUMMARY:
The objective is to evaluate the safety and pharmacokinetic characteristics after co-administration of JW0101 and C2101 and administration of JW0102 in healthy volunteers under fasting conditions

DETAILED DESCRIPTION:
Pharmacokinetic characteristics: Describes the blood concentration statistically by pharmacokinetic blood collection time and treatment group.

Safety: All adverse events are summarized in terms of the number of subjects, expression rate, and number of expressions of adverse reactions by treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Subjects does not meet the Inclusion Criteria

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
AUCt | Day1 0h ~ Day4 72h
  Describes the blood concentration statistically by pharmacokinetic blood collection time and treatment group.
Cmax | Day1 0h ~ Day4 72h
  Describes the blood concentration statistically by pharmacokinetic blood

CONTACTS AND LOCATIONS:
Overall Officials: SeolJu Moon, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Clinical Trial Center, Jeonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No